CLINICAL TRIAL: NCT03601039
Title: Evaluation of Safety and Efficacy of the Absnow Absorbable ASD Closure System For Treating ASD Patients
Brief Title: Safety and Efficacy Study of Absnow Absorbable ASD Closure System For Treating ASD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 42CT（CN）
Record Dates: First submitted 2018-07-06; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Heart Septal Defects, Atrial; Atrial Septal Defect
Keywords: Absnow Absorbable Occluder; ASD Occluder
MeSH Terms: conditions — Heart Septal Defects, Atrial

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Absnow Absorbable ASD Closure System (Experimental): All subjects are implanted with Absnow Absorbable ASD Occluder
  Interventions: Device: Absnow Absorbable ASD Closure System

INTERVENTIONS:
Device: Absnow Absorbable ASD Closure System — the eligible subjects who meet the inclusion criteria should sign the ICF before operation (-30 to 0 day), then receive the Absnow absorbable ASD Closure System implantation. The follow-up time will be set as observation point : the next day after operation, 30-day post-operative , 90-day post-operative, 180-day post-operative, 360-day post-operative, 2 year post-operative, 3 year post-operative, 4 year post-operative and 5 year post-operative. If any AE/SAE occurs during clinical trial, the subjects should be observed till such AE/SAE disappear or stable.

SUMMARY:
The aim of this study is to evaluate the safety and efficacy of Absnow absorbable ASD closure system for treating patients with atrial septal defect.

DETAILED DESCRIPTION:
Atrial Septal Defect (hereinafter referred to as "ASD") is a common congenital heart disease (hereinafter referred to as "CHD"), accounting for about 10% of CHD in children.Initially，ASD was treated by surgical operation. Nowdays transcatheter ASD closure, characterized by minimal invasion, definite curative effect, short recovery period, and no need for cardiopulmonary bypass, provides a new safe and effective therapy for CHD. According to a large number of clinical reports, the use of transcatheter closure devices for ASD closure has a high success rate, good closure effect and low risk of complications.

Absnow absorbable ASD closure system has undergone implantation experiments that implant it into animal (pig) ASD models, with the implantation success rate being 100%. Up to 2 years' observation indicated that the cardiomyocytes and endothelial cells covering the implanted device were not different from those of the control group (nickel-titanium alloy occluder) and were of a great number, and the inflammatory response was remarkably lower than that of the control group. During the observation period, all occluders in the trial did not fall off or were displaced, no evident postoperative complications and therefore, this occluder has the feasibility of local application and system safety.

Absnow absorbable ASD closure system developed by LifeTech Scientific passed the registration inspection of CFDA Shenzhen Medical Device Quality Monitoring and Inspection Center, verifying that this closure system conforms to the product technical specification in mechanical strength, physiochemical properties and biological properties. According to the provisions in Measures for Administration of Medical Device Registration (No. 4 Order) and Regulation on Quality Management of Medical Device Clinical Trial (No. 25) issued by CFDA, this product has the conditions for clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥3 , weight ≥10Kg
* Secundum left-to-right shunt ASD with hemodynamic significance
* Distance from the defect edge to coronary vein sinus, superior and inferior vena cava, pulmonary vein≥5mm and AV valve should be ≥7mm
* The atrial septum length (stretched diameter) should be greater than the diameter of left disk

Exclusion Criteria:

* Patients of primum, venous sinus and coronary sinus ASD
* Patients with atrial septum defect ≥26mm
* Patients with other structural heart disease in addition to ASD
* Patients with complication of obstructive pulmonary arterial hypertension, Eisenmenger syndrome
* Infective endocarditis patients
* Patients with hemolysis or hemorrhagic disease, unhealed ulcer or any taboo about aspirin (except being able to take other anti-platelet agent for consecutive six months) within one month before implantation
* Patients with thrombosis(especially in left atrium or left atrial appendage thrombus) as shown by echocardiography
* Patients with known condition of hypercoagulation status
* Patients ever received heart operation
* Patients allergic to PLLA
* Patients refusing to sign the informed consent form
* Patients with poor compliance on treatment and poor cooperation on follow-up visits
* Patients that are in pregnancy or lactation, or planned for pregnancy or get a positive pregnancy test result during the screening period
* Patients that have participated in any clinical trial that may affect the evaluation of the device in this trial and not completed or withdrawn from the previous clinical trial within 3 months prior to this trial screening period
* The patients considered to be not eligible for this clinical trial by the investigator

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
The successful rate at 30-day post ASD closure operative,which meaning that the TTE or TEE observation shows that residual shunt <5mm at 30-days postoperative. | 30-day post ASD closure operative
  The successful rate at 30-day post ASD closure operative,which meaning that the TTE or TEE observation shows that residual shunt <5mm at 30-days postoperative.
The rate of severe complication during 360-day post ASD closure operative | 360-day post ASD closure operative
  The rate of severe complication during 360-day post ASD closure operative. The severe complication includes all-cause mortality,coronary artery aeroembolism ,cardiac tamponade ,thromboembolism ,occluder dislodgment,repeated migraine, migraine,occluder displacement,mitral regurgitation,heart or aortic root perforation, high degree atrioventricular block and moderate to large residual shunt.

SECONDARY OUTCOMES:
immediate operation success rates | immediate postoperative
  the occluder is successfully implanted which means left and right disks are effectively fixed on left and right sides of atrial septum, respectively and smoothly released without displacement or falling off and the delivery system and the delivery system is successfully withdrawn.
Device-related AE (adverse event) rates | 5 years post operation
  AE refers to adverse medical events occurring during clinical trial no matter if they are device-related
Device-related SAE (serious adverse event) rates | 5 years post operation
  SAE refers to events occurring in the clinical trial that can lead to death or serious health deterioration, including fatal disease or injure, permanent defects of body structure or function, need for hospitalization or prolonging hospitalization time or medial or operation intervention to avoid permanent defects of body structure or body function, fetal distress, fetal death or congenital anomaly, congenital defects.

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - Pan Xiangbin, Beijing, Beijing Municipality
  - Yi Kaijian, Chongqing, Chongqing Municipality
  - Zhang Zhiwei, Guangzhou, Guangdong
  - Yu Bo, Harbin, Heilongjiang
  - Fan Taibing, Zhenzhou, Henan
  - Fang Zhenfei, Changsha, Hunan
  - Kong Xiangqing, Nanjing, Jiangsu
  - Chen Sun, Shanghai, Shanghai Municipality
  - Li Fei, Shanghai, Shanghai Municipality
  - Liu Cong, Shenzhen, Shenzhen
  - Gong Fangqi, Hangzhou, Zhejiang

REFERENCES:
- [Background] Jie Ren. Biodegradable Poly(Lactic Acid): Synthesis, Modification, Processing and Applications. Tsinghua University Press, Beijing and Springer-Verlag Berlin Heidelberg 2010
- [Background] Catia Bastioli. Handbook of Biodegradable Polymers. Rapra Technology Limited Shawbury, Shrewsbury, Shropshire, SY4 4NR, UK.
- [Background] Lakshmi S. Nair, Cato T. Laurencin. Biodegradable polymers as biomaterials. Prog. Polym. Sci. 32 (2007) 762-798.
- [Background] Suuronen R, Pohjonen T, Hietanen J, Lindqvist C. A 5-year in vitro and in vivo study of the biodegradation of polylactide plates. J Oral Maxillofac Surg. 1998 May;56(5):604-14; discussion 614-5. doi: 10.1016/s0278-2391(98)90461-x. PMID 9590343
- [Background] Leenslag JW, Pennings AJ, Bos RR, Rozema FR, Boering G. Resorbable materials of poly(L-lactide). VII. In vivo and in vitro degradation. Biomaterials. 1987 Jul;8(4):311-4. doi: 10.1016/0142-9612(87)90121-9. PMID 3663810